CLINICAL TRIAL: NCT07015398
Title: A Phase 1, Two-Part, Open-Label Drug-Drug Interaction Study to Evaluate the Steady State Pharmacokinetics and Safety Following Co-Administration of Nalbuphine Extended-Release Tablets (NAL ER), and Pirfenidone or Nintedanib in Healthy Adult Subjects
Brief Title: A Study of the Pharmacokinetic Interaction Between Pirfenidone, Nintedanib, and Nalbuphine Extended Release (NAL ER) in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Trevi Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NAL00-105
Record Dates: First submitted 2025-06-03; First posted 2025-06-11 (Actual); Last update posted 2025-10-10 (Actual); Status verified 2025-10

CONDITIONS: Healthy Participants
MeSH Terms: interventions — pirfenidone; nintedanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort A1 - NAL ER + Pirfenidone (Experimental): Participants will receive NAL ER followed by NAL ER co-administered with pirfenidone.
  Interventions: Drug: NAL ER; Drug: Pirfenidone
- Cohort A2 - NAL ER + Nintedanib (Experimental): Participants will receive NAL ER followed by NAL ER co-administered with nintedanib.
  Interventions: Drug: NAL ER; Drug: Nintedanib
- Cohort B1 - Pirfenidone + NAL ER (Experimental): Participants will receive pirfenidone followed by pirfenidone co-administered with NAL ER.
  Interventions: Drug: NAL ER; Drug: Pirfenidone
- Cohort B2 - Nintedanib + NAL ER (Experimental): Participants will receive nintedanib followed by nintedanib co-administered with NAL ER.
  Interventions: Drug: NAL ER; Drug: Nintedanib

INTERVENTIONS:
Drug: NAL ER — Oral tablets
  Other Names: Nalbuphine Extended Release
Drug: Pirfenidone — Oral tablets
  Other Names: ESBRIET®
  Arms: Cohort A1 - NAL ER + Pirfenidone; Cohort B1 - Pirfenidone + NAL ER
Drug: Nintedanib — Oral capsules
  Other Names: OFEV®
  Arms: Cohort A2 - NAL ER + Nintedanib; Cohort B2 - Nintedanib + NAL ER

SUMMARY:
The primary purpose of this study is to evaluate the effect of steady-state NAL ER on the pharmacokinetics (PK) of pirfenidone or nintedanib and the effect of steady-state pirfenidone or nintedanib on the PK of NAL ER in healthy participants.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) ≥ 18.0 and ≤ 30.0 kilogram per meter square (kg/m^2) at Screening.
* Medically healthy with no clinically significant medical history, physical examination, laboratory profiles, vital signs or electrocardiograms (ECGs), as deemed by the principal investigator (PI) or designee.

Exclusion Criteria:

* Positive results for coronavirus infection (COVID-19).
* History or presence of alcohol or drug abuse.
* Positive urine drug or alcohol results.
* Smoker who has used nicotine containing products within the last 3 months.
* History or presence of hypersensitivity or idiosyncratic reaction to the study drugs or related compounds.
* Hemoglobin, absolute neutrophil count, or platelet levels outside of the reference range at Screening.
* History of prolonged QT syndrome or a QTc interval.
* Abnormal liver function at Screening or historical or concurrent liver disease.
* Positive results for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg) or hepatitis C virus (HCV).
* Abnormal Estimated glomerular filtration rate (eGFR).
* History of difficulty donating blood or donation of blood or plasma within 56 days of Screening.
* Participation in another clinical study within 30 days of the baseline visit.

[Note: Other inclusion/exclusion criteria mentioned in the protocol may apply.]

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 132 (Actual)
Dates: Start 2025-06-30 (Actual); Primary Completion 2025-09-12 (Actual); Study Completion 2025-09-26 (Actual)

PRIMARY OUTCOMES:
Maximum Plasma Concentration (Cmax) of NAL ER, Pirfenidone, and Nintedanib | Pre-dose and at multiple timepoints post-dose on Days 1 and 6 for Cohorts A1 and B1; on Days 1 and 8 for Cohort A2; on Days 1 and 7 for Cohort B2
Time to Reach Maximum Observed Concentration (Tmax) of NAL ER, Pirfenidone, and Nintedanib | Pre-dose and at multiple timepoints post-dose on Days 1 and 6 for Cohorts A1 and B1; on Days 1 and 8 for Cohort A2; on Days 1 and 7 for Cohort B2
Area Under the Concentration-Time Curve From Time Zero to Time of Last Measurable Concentration (AUC0-Tlast) of NAL ER, Pirfenidone, and Nintedanib | Pre-dose and at multiple timepoints post-dose on Days 1 and 6 for Cohorts A1 and B1; on Days 1 and 8 for Cohort A2; on Days 1 and 7 for Cohort B2
Area Under the Concentration-Time Curve From Time Zero Extrapolated to Infinity (AUC0-inf) of NAL ER, Pirfenidone, and Nintedanib | Pre-dose and at multiple timepoints post-dose on Days 1 and 6 for Cohorts A1 and B1; on Days 1 and 8 for Cohort A2; on Days 1 and 7 for Cohort B2
Apparent Terminal Rate Constant (λz) of NAL ER, Pirfenidone, and Nintedanib | Pre-dose and at multiple timepoints post-dose on Days 1 and 6 for Cohorts A1 and B1; on Days 1 and 8 for Cohort A2; on Days 1 and 7 for Cohort B2
Apparent Terminal Half-Life (t1/2) of NAL ER, Pirfenidone, and Nintedanib | Pre-dose and at multiple timepoints post-dose on Days 1 and 6 for Cohorts A1 and B1; on Days 1 and 8 for Cohort A2; on Days 1 and 7 for Cohort B2
Apparent Clearance (CL/F) of NAL ER, Pirfenidone, and Nintedanib | Pre-dose and at multiple timepoints post-dose on Days 1 and 6 for Cohorts A1 and B1; on Days 1 and 8 for Cohort A2; on Days 1 and 7 for Cohort B2
Apparent Volume of Distribution (Vz/F) of NAL ER, Pirfenidone, and Nintedanib | Pre-dose and at multiple timepoints post-dose on Days 1 and 6 for Cohorts A1 and B1; on Days 1 and 8 for Cohort A2; on Days 1 and 7 for Cohort B2

SECONDARY OUTCOMES:
Safety and Tolerability as Assessed by Number of Participants With Treatment Emergent Adverse Events (TEAEs) | Up to Day 21
Number of Participants With Clinically Significant Abnormalities in Vital Signs | Up to Day 21

CONTACTS AND LOCATIONS:
Overall Officials: Chief Development Officer, Study Director — Trevi Therapeutics
Locations (1):
- Clinical Pharmacology of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No